CLINICAL TRIAL: NCT02275026
Title: Trajectory of Recovery in the Elderly
Acronym: TORIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Yale University (Other)
Responsible Party: Principal Investigator, Joshua Mincer, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO 13-0359; 1R01AG046634 (NIH)
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Delayed Emergence From Anesthesia; Postoperative Delirium; Postoperative Cognitive Dysfunction
Keywords: General Anesthesia, Postoperative Delirium, Recovery
MeSH Terms: conditions — Delayed Emergence from Anesthesia; Emergence Delirium; Postoperative Cognitive Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Functional magnetic resonance imaging (Experimental): Magnetic resonance images will be acquired on a 3 Tesla scanner (Skyra, Siemens, Erlangen, Germany) with a 20 channel receiver coil.
  Interventions: Procedure: Functional magnetic resonance imaging

INTERVENTIONS:
Procedure: Functional magnetic resonance imaging — Diffusion tensor imaging
  Other Names: fMRI

SUMMARY:
The purpose of this study is to understand how elderly individuals regain their cognitive skills following general anesthesia. The investigators will compare an age stratified group of volunteers who will be evaluated with a series of cognitive tests and a functional MRI. The participants will then be administered general anesthesia for two hours. The investigators will then assess the participants using state of the art tools to determine when participants return to their cognitive baseline.

DETAILED DESCRIPTION:
Elderly patients undergoing anesthesia and surgery frequently suffer from postoperative cognitive dysfunction (POCD) and postoperative delirium (PD). The cause of these entities is unknown. It is unclear what part anesthetics play in the development of POCD and PD. The investigators hypothesize that elderly patient's cognitive capacities recover more slowly after receiving general anesthesia, perhaps because they have more limited cognitive reserve. A more prolonged recovery would confound diagnoses of POCD and PD and potentially puts patients who are discharged on the day of surgery at risk of not understanding postoperative instructions. The trajectory of postoperative cognitive recovery has never been explored and elderly participants have been explicitly not included in any type of emergence research. To explore this vital area the investigators propose to study young and elderly volunteers with a combination of two state of the art neuropsychological tests (Postoperative Quality of Recovery Scale and the NIH Toolbox) and functional magnetic resonance imaging. Starting from baseline, the investigators will determine multiple cognitive domains and resting state networks, treat the participants with general anesthesia for two hours while continuing to examine network activity, and then explore the recovery of the cognitive domains and alterations in functional networks using both the PQRS and the NIH Toolbox Cognitive Measures. Participants will be evaluated at 1 month, 6 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 40-80 years old
* American Society of Anesthesiologists (ASA) Physical Status I or II (i.e. Individuals with minimal disease burden)
* Capable and willing to consent

Exclusion Criteria:

* Airway assessment as potentially difficult (Mallampati III or greater)
* Allergies or hypersensitivity to drug or class
* Chronic Inflammatory conditions such a lupus or system rheumatoid arthritis (arthritis limited to 1 or 2 joints will be acceptable)
* Patients with diabetes mellitus
* Patients with a recent illness (within the last 2 weeks)
* Patients with severe visual or auditory disorder/handicaps
* English illiteracy
* Pregnancy
* Participants not expected to be able to complete the postoperative tests
* History of malignant hyperthermia
* Nursing mothers
* Body Mass Index > 30
* Patients with significant metal implants in body
* Current use of cocaine or opiates
* Current smokers

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2015-07; Primary Completion 2020-04-22 (Actual); Study Completion 2020-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Mincer, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Baxter MG, Mincer JS, Brallier JW, Schwartz A, Ahn H, Nir T, McCormick PJ, Ismail M, Sewell M, Allore HG, Ramsey CM, Sano M, Deiner SG. Cognitive Recovery by Decade in Healthy 40- to 80-Year-Old Volunteers After Anesthesia Without Surgery. Anesth Analg. 2022 Feb 1;134(2):389-399. doi: 10.1213/ANE.0000000000005824. PMID 34889804
- [Derived] Nir T, Raizman R, Meningher I, Jacob Y, Huang KH, Schwartz AE, Brallier JW, Ahn H, Kundu P, Tang CY, Delman BN, McCormick PJ, Scarpa J, Sano M, Deiner SG, Livny A, Baxter MG, Mincer JS. Lateralisation of subcortical functional connectivity during and after general anaesthesia. Br J Anaesth. 2022 Jan;128(1):65-76. doi: 10.1016/j.bja.2021.08.033. Epub 2021 Nov 19. PMID 34802696
- [Derived] Nir T, Jacob Y, Huang KH, Schwartz AE, Brallier JW, Ahn H, Kundu P, Tang CY, Delman BN, McCormick PJ, Sano M, Deiner S, Baxter MG, Mincer JS. Resting-state functional connectivity in early postanaesthesia recovery is characterised by globally reduced anticorrelations. Br J Anaesth. 2020 Oct;125(4):529-538. doi: 10.1016/j.bja.2020.06.058. Epub 2020 Aug 14. PMID 32800503
- [Derived] Deiner S, Baxter MG, Mincer JS, Sano M, Hall J, Mohammed I, O'Bryant S, Zetterberg H, Blennow K, Eckenhoff R. Human plasma biomarker responses to inhalational general anaesthesia without surgery. Br J Anaesth. 2020 Sep;125(3):282-290. doi: 10.1016/j.bja.2020.04.085. Epub 2020 Jun 11. PMID 32536445
- [Derived] Mincer JS, Baxter MG, McCormick PJ, Sano M, Schwartz AE, Brallier JW, Allore HG, Delman BN, Sewell MC, Kundu P, Tang CY, Sanchez A, Deiner SG. Delineating the Trajectory of Cognitive Recovery From General Anesthesia in Older Adults: Design and Rationale of the TORIE (Trajectory of Recovery in the Elderly) Project. Anesth Analg. 2018 May;126(5):1675-1683. doi: 10.1213/ANE.0000000000002427. PMID 28891911

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was completed in May 2019.
Groups:
- Functional Magnetic Resonance Imaging: Magnetic resonance images acquired on a 3 Tesla scanner (Skyra, Siemens, Erlangen, Germany) with a 20 channel receiver coil.
  Functional magnetic resonance imaging: Diffusion tensor imaging
Period: Overall Study
Arm/Group | Functional Magnetic Resonance Imaging
Started | 104
Completed | 71
Not Completed | 33
Not completed — Ineligible after cognitive baseline testing | 11
Not completed — Withdrawal by Subject | 4
Not completed — Ineligible due to medical history | 13
Not completed — MRI malfunction precluded testing | 1
Not completed — Ineligible after MRI findings | 1
Not completed — Lost to Follow-up | 2
Not completed — Scanner failure | 1

BASELINE CHARACTERISTICS:
Population: Participants who completed Day 1 Scan
Arm/Group | Functional Magnetic Resonance Imaging
Number analyzed (Participants) | 72
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [48.5 to 69.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 63
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 31
  White | 34
  More than one race | 3
  Unknown or Not Reported | 1
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 26.5 [24.3 to 28.4]
ASA Physical Status [Count of Participants; unit: Participants] — American Society of Anesthesiologists Physical Status Classification System. Classification 1- 6, higher score indicates poorer health outcomes.
  Participants
    1 - A normal healthy patient | 57
    2 - A patient with mild systemic disease without substantive functional limitations | 15
Disease History [Count of Participants; unit: Participants]
  Hypertension | 3
  Asthma | 1
  Malignancy (any) | 7
Number of medications on initial assessment [Count of Participants; unit: Participants]
  0 | 61
  1 | 4
  2 | 6
  3+ | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Recovered on Postoperative Quality of Recovery Scale (PQRS)
Description: Cognitive Function using scales of the PQRS to test whether age is associated with the time of return to baseline cognitive function. The PQRS is a brief measurement tool to assess multiple domains of recovery, including cognition, over time. It is scored as recovered / not recovered based on level of performance, within a certain tolerance range, relative to preoperative (baseline) performance - before the general anesthesia / MRI scanning session. Postoperative Quality of Recovery Cognitive Scale at each study timepoint by age decade. Postoperative Quality of Recovery Cognitive
Time Frame: 15 min, 60 min, 1 day, 3 days, 7 days, 30 days, 6 months
Population: Scale could not be determined for 2 participants (1 in the 40-49 year age decade, one in the 70-80 year age decade).
Measure: Count of Participants; unit: Participants
Groups:
- Age Decade 40-49; Age Decade 50-59; Age Decade 60-69; Age Decade 70-80: Groups divided by age decade
Arm/Group | Age Decade 40-49 | Age Decade 50-59 | Age Decade 60-69 | Age Decade 70-80
Number analyzed (Participants) | 19 | 19 | 13 | 18
Participants
  at 15 min | 3 | 5 | 1 | 3
  at 60 min | 8 | 11 | 8 | 9
  1 day | 17 | 18 | 12 | 16
  3 days | 18 | 19 | 12 | 17
  7 days | 18 | 19 | 12 | 17
  30 days | 18 | 19 | 12 | 18
  6 months | 19 | 19 | 13 | 18

2. Secondary Outcome: Change in NIH Tool Box Composite
Description: NIH Toolbox Cognitive Battery is a multidimensional set of brief measures assessing cognitive (as well as emotional, motor and sensory) function. There is no score range, but mean score is 100 with standard deviation 15. A score at or near 100 indicates average ability compared with others. Scores around 115 suggest above-average ability. Scores around 130 suggest superior ability (in the top 2 percent nationally). A score around 85 suggests below-average ability. A score in the range of 70 or below suggests significant impairment.
Time Frame: Baseline, 1 day, 7 days, 30 days
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Age Decade 40-49 | Age Decade 50-59 | Age Decade 60-69 | Age Decade 70-80
Number analyzed (Participants) | 20 | 19 | 13 | 19
score on a scale
  Baseline | 48.1 [45.3 to 51.0] | 53.3 [50.3 to 56.3] | 50.1 [16.5 to 53.7] | 54 [51.0 to 56.9]
  1 day | 52.2 [49.4 to 55.1] | 57.2 [54.2 to 60.2] | 53.2 [49.6 to 56.8] | 57.4 [54.4 to 60.3]
  7 days | 54.8 [52 to 57.7] | 59.4 [56.4 to 62.4] | 54.6 [50.9 to 58.2] | 54.4 [50.7 to 58.1]
  30 days | 54.5 [51.6 to 57.4] | 59.5 [56.5 to 62.5] | 54.4 [50.7 to 58.1] | 59.6 [56.7 to 62.6]

ADVERSE EVENTS:
Time Frame: 30 days
Description: According to Michigan Awareness Classification Instrument
Arm/Group | Functional Magnetic Resonance Imaging
All-Cause Mortality (participants affected / at risk) | 0/72
Serious Adverse Events (participants affected / at risk) | 0/72
Other Adverse Events (participants affected / at risk) | 4/72
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Functional Magnetic Resonance Imaging (N=72)
Sore Throat (Injury, poisoning and procedural complications) | 1
Nausea (Gastrointestinal disorders) | 1
Eye discomfort (Eye disorders) | 1
Lingual nerve compression injury (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/26/NCT02275026/Prot_000.pdf
  • Statistical Analysis Plan (2013-10-31): https://cdn.clinicaltrials.gov/large-docs/26/NCT02275026/SAP_001.pdf